CLINICAL TRIAL: NCT03437291
Title: Comparison Between the Role of Transabdominal Ultrasound Versus Transvaginal Ultrasound in Evaluation of Placental Invasion in Cases of Placenta Previa Anterior Wall With Previous Uterine Scar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 27
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abnormal placental invasion: patients had placenta previa with histopathologically confirmed abnormal invasion with all three grades i.e. accreta, increta and percreta,
  Interventions: Procedure: Cesarean section; Device: Transabdominal ultrasound; Device: Transvaginal ultrasound
- Normal placenta: patients had placenta previa with no abnormal invasion
  Interventions: Procedure: Cesarean section; Device: Transabdominal ultrasound; Device: Transvaginal ultrasound

INTERVENTIONS:
Procedure: Cesarean section — Lower segment CS with evaluation of Placental site, spontaneous separation, placental invasion into the bladder and other surrounding organs, Uterotonic administration, Bladder , ureteric or bowel injury, blood loss and blood transfusion
  Other Names: lower segment cesarean section
Device: Transabdominal ultrasound — loss of clear zone, Abnormal placental lacunae, Bladder wall interruption, Myometrial thinning, Placental bulge, Focal exophytic mass
  Other Names: 2D ultrasound system equipped with a 4-8-MHz trans-abdominal transducer
Device: Transvaginal ultrasound — loss of clear zone, Abnormal placental lacunae, Bladder wall interruption, Myometrial thinning, Placental bulge, Focal exophytic mass
  Other Names: 2D ultrasound system equipped with a 12 MHz transvaginal transducer

SUMMARY:
Objective:

To compare between the role of Transabdominal ultrasound versus Transvaginal ultrasound in evaluation of placental invasion in cases of placenta previa anterior wall with previous uterine scar applying the unified ultrasonographic descriptors suggested by the European working group on abnormally invasive placenta "EW-AIP' Also to evaluate the sensitivity and specificity of each criterion by comparing them with the final outcome of pregnancy Fifty pregnant women with persistent placenta previa (after 28 weeks' gestation) were prospectively enrolled into this study. Both transabdominal and transvaginal ultrasound were performed by two different operators who were blinded to the results of each other.

the placenta was studied as regarding the exact loacalization and the unified descriptors were applied and evaluated by TAS and TVS.

The ultrasound findings were analyzed with reference to the final diagnosis made during Cesarean delivery and histopathological examination

DETAILED DESCRIPTION:
Definitive diagnosis of Abnormally Invasive Placenta was made at delivery when the myometrium was seen to be invaded by the placenta, and the pathological examination of the removed uterus showed the villi attached to the myometrium without intervening decidua (accreta), invading into the myometrium (increta) or reaching the serosa (percreta).

-Complete imaging using all diagnostic techniques (gray-scale, color Doppler) by both transabdominal and transvaginal by two expert operators, then an offline analysis of the acquired images & volumes was done Ultrasound examination was performed using a 2D ultrasound system equipped with a 4-8-MHz trans-abdominal transducer and a 12 MHz transvaginal transducer The transvaginal ultrasound was performed by a highly experienced operator whereas the transabdominal ultrasound was performed by a less experienced one and both were blinded from the results of each other Placenta was examined while the bladder was partially full about 300 ml for adequate visualization and precise localization

The Examined placenta is considered to be suspicious of abnormal invasion in case of having one or more of the unified descriptors described by the European working Group on Abnormally Invasive Placenta "EW-AIP":

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the reproductive age group (18 - 45) diagnosed persistent placenta previa anterior wall after 28 weeks of gestation , with history of previous Caesarian Section and/or any other type of uterine surgeries

Exclusion Criteria:

* Placenta previa posterior wall
* unscarred uterus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women in the reproductive age group (18 - 45) diagnosed persistent placenta previa anterior wall after 28 weeks of gestation , with history of previous Caesarian Section and/or any other type of uterine surgeries
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
abnormal placental invasion | At time of cesarean section
  detection of abnormally invsive placenta at histopathological examination

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided